CLINICAL TRIAL: NCT02059213
Title: A Randomized Phase II Study of Androgen Deprivation Therapy With or Without Palbociclib in RB-Positive Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: A Phase II Study of Androgen Deprivation Therapy With or Without Palbociclib in RB-Positive Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: University of Utah (Other); Vanderbilt-Ingram Cancer Center (Other); Johns Hopkins University (Other); Thomas Jefferson University (Other); Washington University School of Medicine (Other); Northwestern University (Other); City of Hope Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.117; HUM00082715 (Other: University of Michigan)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — palbociclib; bicalutamide; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADT Alone (Active Comparator): Androgen Deprivation Therapy (ADT): Bicalutamide (an active non-steroidal antiandrogen; 50mg taken daily by mouth) and Zoladex (LHRH agonist administered by injection), or Lupron Depot (LHRH agonist, administered by injection).
  Interventions: Drug: Bicalutamide; Drug: Zoladex; Drug: Lupron Depot
- ADT + Ibrance® (Experimental): Ibrance® (125mg taken daily by mouth days 1-21 of a 28 day cycle) in addition to Androgen Deprivation Therapy (ADT): Bicalutamide (an active non-steroidal antiandrogen; 50mg taken daily by mouth) and Zoladex (LHRH agonist administered by injection), or Lupron Depot (LHRH agonist, administered by injection).
  Interventions: Drug: Ibrance; Drug: Bicalutamide; Drug: Zoladex; Drug: Lupron Depot

INTERVENTIONS:
Drug: Ibrance
  Other Names: PD 0332991; Palbociclib
  Arms: ADT + Ibrance®
Drug: Bicalutamide
  Other Names: Casodex
Drug: Zoladex
  Other Names: Goserelin acetate implant
Drug: Lupron Depot
  Other Names: Leuprolide

SUMMARY:
This study will look at the effect of adding the drug Palbociclib to CAD (Combined Androgen Deprivation) therapy in patients with RB (Retinoblastoma Protein) positive hormone sensitive prostate cancer.

The investigators hypothesize that the addition of Palbociclib to initial ADT (Androgen Deprivation Therapy) in patients with newly metastatic RB-positive prostate cancer may significantly increase the efficacy of ADT.

DETAILED DESCRIPTION:
Patients will undergo exams, tests, and procedures to determine if they are eligible to participate. Subjects will be randomized to one of two groups. Patients randomized to Arm 1 - Patients will receive the LHRH agonist every 3 months. Patients will also take 50 mg. of bicalutamide by mouth every day. Bicalutamide comes in tablet form. This arm is broken down into periods of time called cycles, starting with cycle 1 then cycle 2, and so on.Each cycle is 28 days long. If randomized to Arm 2 - Patients will receive the LHRH agonist every 3 months. Patients will also take 50 mg. of bicalutamide by mouth every day. Patients will also take 125 mg. of Ibrance® daily for 21 days, and then will stop taking Ibrance® for 7 days. Patients will then begin taking Ibrance® again after 7 days off. Patients will keep repeating this cycle every 28 days. When the patient starts the first 28 day cycle that will be cycle 1, then cycle 2, and so on. During each cycle the patient will come in for routine and research tests and procedures for patient safety, to see how patients are doing, and for research purposes. The researchers will ask patients to complete a drug diary to track bicalutamide and Ibrance® administration. The total time of study participation depends on how a patient responds to the study medications. Patients may be on the study for a short period of time, such as a week, or for a longer period of time, such as a few years. Patients may continue on study treatment until one of the following: cancer progresses (gets worse); another illness or condition develops that prevents study participation; unacceptable side effects occur; drug is delayed more than 4 weeks; patient withdraws consent; the study doctor thinks the patient should stop; the patient does not follow researcher's instructions; the study is cancelled.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologic diagnosis of prostate cancer.
* Have hormone-sensitive metastatic disease (M1) as evidenced by soft tissue and/or bony metastases.
* Patients may either be untreated for their newly diagnosed metastatic disease (preferred as much as possible) or have started androgen deprivation therapy. Patients who have started androgen deprivation therapy for the treatment of their newly diagnosed metastatic disease are eligible as long as the duration of treatment is less than or equal to 2 weeks (14days) prior to registration. The start date of androgen deprivation is considered the day the patient first received an injection of a LHRH agonist/antagonist (or orchiectomy), not the date when an oral antiandrogen started.
* Patients must have a minimum PSA (Prostate-Specific Antigen) ≥ 5 ng/mL within 60 days of registration or prior to the initiation of androgen deprivation for patients who have started androgen deprivation therapy.
* Agree to undergo a biopsy of at least one metastatic site for RB (Retinoblastoma Protein) status evaluation. Adequate metastatic tissue from prior biopsy/resection can be used if available in lieu of a biopsy.
* ECOG performance status of 0-2 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death).
* Patients may have received prior neoadjuvant and/or adjuvant hormonal therapy, for non-metastatic disease but it must not have lasted for more than 36 months. At least 12 months must have elapsed since completion of androgen deprivation therapy in the neoadjuvant and/or adjuvant setting.
* Within 14 days prior to registration patients must have adequate organ and marrow function: White Blood Cell (WBC) count ≥ 3,000/μl, Absolute Neutrophil Count (ANC) ≥ 1,500/μl, Platelet Count ≥ 100,000/μl, Serum Creatinine ≥1.5 x the institutional upper limits of normal or corrected creatinine clearance of ≥ 50 mg/ml/hr/1.73 m2 BSA (Body Surface Area), Bilirubin within the institutional limits of normal, AST (Aspartate Aminotransferase) ≤ 2 x upper limits of normal, ALT (Alanine Aminotransferase) ≤ 2 x upper limits of normal.
* Patients must be able to take oral medication without crushing, dissolving or chewing tablets.
* Patients may have received prior radiation therapy or surgery. However, at least 14 days must have elapsed since completion of radiation therapy or surgery and patient must have only grade 2 or less adverse effects at the time of registration.
* Patients must agree to use highly effective contraception during treatment and for a period of 90 days after ending treatment with PD 0332991.
* Ability to understand and the willingness to sign a written informed consent document that is approved by an institutional review board.

Exclusion Criteria:

* Patients who have received androgen deprivation therapy for greater than 14 days (LHRH-agonist or antagonist) for the treatment of their newly diagnosed metastatic disease prior to enrollment are not eligible for this study.
* Patients who are currently being treated with strong CYP3A4 inhibitors (e.g., amprenavir, fosamprenavir, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, voriconazole, and grapefruit) or strong inducers (e.g., carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, primidone, rifabutin, rifampin, rifapentine and St. John's wort) must either discontinue these drugs or are ineligible.
* Patients must refrain from the use of proton pump inhibitors. If needed, alternative antacid therapies may be used including H2-receptor antagonists, and locally acting antacids.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible. Patients are not considered to have a "currently active" malignancy if they have completed all therapy and are now considered without evidence of disease for 1 year.
* HIV-positive patients on combination antiretroviral therapy are ineligible .

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-06; Primary Completion 2017-09-09 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, MD, FACP, FASCO, Principal Investigator — University of Michigan Comprehensive Cancer Center and Northwestern University
Locations (8):
- United States (8):
  - City of Hope Cancer Center, Duarte, California
  - Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Palmbos PL, Daignault-Newton S, Tomlins SA, Agarwal N, Twardowski P, Morgans AK, Kelly WK, Arora VK, Antonarakis ES, Siddiqui J, Jacobson JA, Davenport MS, Robinson DR, Chinnaiyan AM, Knudsen KE, Hussain M. A Randomized Phase II Study of Androgen Deprivation Therapy with or without Palbociclib in RB-positive Metastatic Hormone-Sensitive Prostate Cancer. Clin Cancer Res. 2021 Jun 1;27(11):3017-3027. doi: 10.1158/1078-0432.CCR-21-0024. Epub 2021 Mar 16. PMID 33727260

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 72 patients were enrolled to the trial. Seven patients did not have adequate tissue for testing retinoblastoma status. Two patients tested negative for retinoblastoma and one patient was found to have small cell metastasis and not adenocarcinoma. 62 patients were randomized.
Period: Overall Study
Arm/Group | ADT Alone | ADT + Ibrance®
Started | 20 | 42
Initiated Treatment | 20 | 40
Completed | 20 | 40
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: 62 out of 72 patients enrolled had adequate tissue for RB assessment and retained RB expression. (60 patients initiated treatment.)
Groups:
- Total: Total of all reporting groups
Arm/Group | ADT Alone | ADT + Ibrance® | Total
Number analyzed (Participants) | 20 | 42 | 62
Age, Continuous [Median (Full Range); unit: years] | 67.5 [44 to 81] | 67.5 [47 to 87] | 67.5 [44 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 42 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 16 | 39 | 55
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve a PSA ≤ 4ng/mL After Seven Months of Protocol Treatment in Each Arm
Description: The primary analysis will be assessment of the proportion of patients who achieve a (Prostate-specific antigen) PSA < 4ng/mL after seven months of protocol treatment in each arm.
Time Frame: 28 weeks
Population: 72 patients were enrolled to the trial. Seven patients did not have adequate tissue for testing retinoblastoma status. Two patients tested negative for retinoblastoma and one patient was found to have small cell metastasis and not adenocarcinoma. 62 patients were randomized. 60 randomized patients initiated therapy on trial.
Measure: Count of Participants; unit: Participants
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
Participants | 16 | 32
Statistical Analysis 1: Comparison: ADT Alone vs ADT + Ibrance®; With 20 patients treated with ADT and 40 treated with ADT + palbociclib there is a 64.2% power to detect a 20% difference in proportions with a one-sided type I error of 0.10 using the mid p-value method of the Fisher's exact test; Test type: Superiority; p = 0.87, Fisher Exact; Mid P-value

2. Secondary Outcome: Number of Participants With Grade >=3 Adverse Events That Are Possibly, Probably or Definitely Related to Study Treatment
Description: Grade >=3 adverse events that are possibly, probably or definitely related to study treatment, reported by number of participants affected in each arm
Time Frame: Up to 54 months
Measure: Number; unit: participants
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
participants | 0 | 23

3. Secondary Outcome: Duration of Therapy
Description: Duration of therapy will be reported to describe tolerability within each arm.
Time Frame: Up to 54 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
months | 22.4 (13.1) | 22.0 (13.8)
Statistical Analysis 1: Comparison: ADT Alone vs ADT + Ibrance®; Test type: Superiority; p = 0.92, t-test, 2 sided

4. Secondary Outcome: Proportion of Patients Who Achieve Undetectable PSA (<0.2ng/mL)
Time Frame: Up to 54 months
Measure: Count of Participants; unit: Participants
Groups:
- ADT Alone: Androgen Deprivation Therapy (ADT): Bicalutamide (an active non-steroidal antiandrogen; 50mg taken daily by mouth) and Zoladex (LHRH agonist administered by injection), or Lupron Depot (LHRH agonist, administered by injection).
  Bicalutamide
  Zoladex
  Lupron Depot
- ADT + Ibrance®: Ibrance® (125mg taken daily by mouth days 1-21 of a 28 day cycle) in addition to Androgen Deprivation Therapy (ADT): Bicalutamide (an active non-steroidal antiandrogen; 50mg taken daily by mouth) and Zoladex (LHRH agonist administered by injection), or Lupron Depot (LHRH agonist, administered by injection).
  Ibrance
  Bicalutamide
  Zoladex
  Lupron Depot
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
Participants | 13 | 22
Statistical Analysis 1: Comparison: ADT Alone vs ADT + Ibrance®; Test type: Superiority; p = 0.50, Fisher Exact; Mid p-value

5. Secondary Outcome: Biochemical Progression-free Survival Rate
Description: 12-month biochemical progression-free survival rate will begin from treatment start until the event of biochemical (PSA) progression or death, whichever occurs first. Described by arm using Kaplan-Meier methods.
Time Frame: Up to 54 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
percentage of participants
  12-month | 74.7 [49.4 to 88.6] | 76.5 [59.6 to 87]
  26-month (time of last event in Arm 1) | 45.8 [22.4 to 66.6] | 59.4 [41.7 to 73.3]
  43-month (time of last event in Arm 2) | 45.8 [22.4 to 66.6] | 33.9 [8.9 to 61.7]
Statistical Analysis 1: Comparison: ADT Alone vs ADT + Ibrance®; Test type: Superiority; p = 0.72, Log Rank

6. Secondary Outcome: Clinical Progression-free Survival Rate
Description: 12-month clinical progression-free survival rate will begin from treatment start until the event of biochemical (PSA) progression or death, whichever occurs first. Described by arm using Kaplan-Meier methods.
Time Frame: Up to 54 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
percentage of participants
  12-month | 77.7 [51.1 to 91] | 83.8 [67.4 to 92.4]
  22-month (time of last event in Arm 1) | 64.8 [37.5 to 82.5] | 77.7 [60.2 to 88.2]
  32-month (time of last event in Arm 2) | 64.8 [37.5 to 82.5] | 58.5 [33.9 to 76.6]
Statistical Analysis 1: Comparison: ADT Alone vs ADT + Ibrance®; Test type: Superiority; p = 0.76, Log Rank

7. Secondary Outcome: Frequency of Dose Modification
Description: Dose modifications will be reported to describe tolerability for arm 2 only (Ibrance®)
Time Frame: Up to 54 months
Measure: Number; unit: participants
Arm/Group | ADT + Ibrance®
Number analyzed (Participants) | 40
participants
  No Dose Reduction (Palbociclib 125mg/day) | 28
  1 Dose Reduction, to Palbociclib 100mg/day | 5
  2 Dose Reductions, to Palbociclib 75mg/day | 7

8. Secondary Outcome: Frequency of Treatment Delay
Description: Treatment delays will be reported to describe tolerability within each arm.
Time Frame: Up to 54 months
Measure: Number; unit: participants
Arm/Group | ADT Alone | ADT + Ibrance®
Number analyzed (Participants) | 20 | 40
participants
  No Treatment delay of Bicalutamide | 19 | 35
  Treatment Delay of Bicalutamide | 1 | 5
  No Treatment Delay of Palbociclib | 0 | 21
  Treatment Delay of Palbociclib | 0 | 19

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected up to 44 months.
Arm/Group | ADT Alone | ADT + Ibrance®
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/40
Serious Adverse Events (participants affected / at risk) | 5/20 | 7/40
Other Adverse Events (participants affected / at risk) | 20/20 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADT Alone (N=20) | ADT + Ibrance® (N=40)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADT Alone (N=20) | ADT + Ibrance® (N=40)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 13 (23)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) | 3 (5)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1) | 3 (4)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 6 (6)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 14 (18)
Dental caries (Gastrointestinal disorders) | 1 (1) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 10 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2) | 8 (8)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 9 (13)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 5 (17)
Chills (General disorders) | 0 (0) | 5 (5)
Edema limbs (General disorders) | 7 (8) | 9 (11)
Fatigue (General disorders) | 12 (16) | 23 (29)
Fever (General disorders) | 1 (2) | 0 (0)
Flu like symptoms (General disorders) | 3 (6) | 6 (10)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (3) | 8 (10)
Injection site reaction (General disorders) | 0 (0) | 3 (3)
Irritability (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 4 (7) | 12 (17)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (5) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 9 (14)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 5 (7)
Alkaline phosphatase increased (Investigations) | 1 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 6 (9)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (5) | 3 (6)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 2 (2)
Investigations - Other (Investigations) | 2 (2) | 3 (4)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 6 (12)
Neutrophil count decreased (Investigations) | 0 (0) | 25 (96)
Platelet count decreased (Investigations) | 0 (0) | 14 (29)
Weight gain (Investigations) | 6 (12) | 7 (10)
Weight loss (Investigations) | 2 (2) | 3 (6)
White blood cell decreased (Investigations) | 1 (1) | 19 (65)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (13) | 15 (36)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5) | 7 (11)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 9 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (6) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (3)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 9 (13)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (5)
Headache (Nervous system disorders) | 2 (2) | 6 (8)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (5) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 6 (7)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (4)
Depression (Psychiatric disorders) | 3 (3) | 8 (10)
Insomnia (Psychiatric disorders) | 4 (4) | 9 (9)
Libido decreased (Psychiatric disorders) | 2 (2) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 3 (4) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (3) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 7 (7)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (2) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Gynecomastia (Reproductive system and breast disorders) | 4 (4) | 8 (8)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 6 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 16 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (7)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (6) | 10 (13)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 16 (19) | 31 (36)
Hypertension (Vascular disorders) | 2 (2) | 8 (17)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT02059213/Prot_SAP_000.pdf